CLINICAL TRIAL: NCT06160661
Title: Radiographic Assessment of Three Dimensional Mandibular Position Using Splint-less Patient Specific Implant Following Bilateral Sagittal Split Osteotomy
Brief Title: Radiographic Assessment of Three Dimensional Mandibular Position Using Splint-less Patient Specific Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abanoub Fayez Aziz, PhD candidate of oral and maxillofacial surgery , principal investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: FDASU-Rec ID032243
Record Dates: First submitted 2023-11-03; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Abnormality of Facial Skeleton

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm study (Experimental): The purpose of this study was to assess the accuracy of a splint-less approach for mandibular jaw orthognathic surgery. This approach utilized a personalized orthognathic surgical guide (POSG) system, which comprised a set of cutting guides and 3D printed custom titanium fixation plates for bilateral sagittal split osteotomies (BSSOs).
  The cutting guides were first used to predrill screw holes and guide osteotomies. The custom plates were then used to reposition and stabilize the bony segments as planned, without the use of surgical splints or any additional tool such as surgical navigation
  Interventions: Device: mandibular saggital split osteotomy

INTERVENTIONS:
Device: mandibular saggital split osteotomy — orthognathic surgery

SUMMARY:
The purpose of this study was to assess the accuracy of a splint-less approach for mandibular jaw orthognathic surgery. This approach utilized a personalized orthognathic surgical guide (POSG) system, which comprised a set of cutting guides and 3D printed custom titanium fixation plates for bilateral sagittal split osteotomies (BSSOs).

The cutting guides were first used to predrill screw holes and guide osteotomies.

The custom plates were then used to reposition and stabilize the bony segments as planned, without the use of surgical splints or any additional tool such as surgical navigation

DETAILED DESCRIPTION:
Surgical technique:

The buccal bony surface of the mandible was exposed as a routine sagittal split osteotomy. First, the mandibular cutting guide was installed using the tooth-borne splint portion of the guide.

Second, the lower portion of the guide was temporarily fixed with titanium screws through the designed screw holes on the guide. The planned margins for vertical osteotomy/ ostectomy were then marked by a pencil.

Once the cutting guide was removed, the sagittal split osteotomy was completed as usual. Finally, the distal and proximal segments were fixed together using the custom plates and screw holes that were used by the cutting guide.

Accuracy of preoperative surgical planning, and validation of the use of patient specific implants (PSI) in bilateral sagittal split osteotomy (BSSO) by comparing the planned outcomes to the actual postoperative outcomes by two methos.

A)Evaluation the discrepancy between planned and obtained post-operative position of the mandibular plates, rami, and occlusion by analyzing the discrepancies in terms of rotation (roll, pitch and yaw) and translation (antero-posterior, lateral and vertical). These movements were determined by incorporating the segments in homologous bounding-boxes, aligning the planned model to the post-op result colorimetric map inspection.

B) Measurements of the linear differences between the planned and postoperative positions of the mandibular midlines, the chin, and the gonial angle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from skeletal deformity requiring mandibular orthognathic surgery (Bilateral sagittal splitting osteotomy).
2. Patients should be free from any systemic disease that may affect normal bone healing and predictable outcome.

Exclusion Criteria:

1. Patients with metabolic bone disease that affects bone healing.
2. Intra-bony lesions that may affect the osteotomy healing.
3. Patients with history of radiotherapy on the head and neck region

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
device feasibility and eligibility for use of PSI | 1 week postoperative
  The primary outcome of this study is to assess the accuracy of preoperative surgical planning, and validation feasibility of the use of patient specific implants (PSI) in bilateral sagittal split osteotomy (BSSO) by comparing the planned outcomes to the actual postoperative outcomes by two measurement tools (MIMICS software, and DICOM file of pre and post operative CT) . By using software we can superimpose the DICOM files of CT and linear differences in millimetres between fixed points in CT can be obtained to assess the accuracy of the outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No